CLINICAL TRIAL: NCT06213935
Title: Preoperative Oral Midodrine Versus Intraoperative Intravenous Norepinephrine in Preventing Post-spinal Anesthesia Hypotension in Cesarean Section: A Prospective Double-blind Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Andrew Ramsis Khalafallah, Resident of Anesthesia,Intensive Care and Pain control department, Sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med-23-12-01MS
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Post Spinal Anesthesia Hypotension
MeSH Terms: interventions — Norepinephrine; Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): will receive a norepinephrine bolus at 0.05 μg/kg, followed by norepinephrine infusion at a rate of 0.05 μg/kg.min
  Interventions: Drug: Norepinephrine
- Group B (Active Comparator): will receive 10 mg tablets of midodrine 1 hour before spinal anesthesia.
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Norepinephrine — after spinal anesthesia, norepinephrine will be injected intravenous as bolus at 0.05 μg/kg, followed by norepinephrine infusion at a rate of 0.05 μg/kg.min to prevent post spinal hypotension
  Arms: group A
Drug: Midodrine — 10 mg tablets of midodrine 1 hour before spinal anesthesia to prevent post spinal anesthesia hypotension
  Arms: Group B

SUMMARY:
Neuraxial blockade such as spinal anaesthesia can cause severe hypotension due to pharmacological sympathectomy resulting in potential deleterious consequences for the patient, Prevention of this spinal anaesthesia induced hypotension is of utmost importance, Techniques currently in use for preventing hypotension include intravenous fluid prehydration, sympathomimetic drugs, and physical methods such as positioning and leg compression.

Midodrine is an orally active α-adrenergic agonist ,Used in clinical management of patients with orthostatic hypotension or hypotension secondary to other clinical conditions or drug therapies. Midodrine is almost completely absorbed after oral administration and undergoes enzymatic hydrolysis to form its pharmacologically active metabolite, de-glymidodrine , causes venous and arterial vasoconstriction through stimulation of α1- receptors located in the vasculature, However ,Midodrine may cause several side effects as chills ,numbness , tingling ,paresthesia ,polyuria ,dysuria and headache.

On the other hand, Norepinephrine is a vasoconstrictor that predominantly stimulates α1 receptors to cause peripheral vasoconstriction and increase blood pressure. It also has some β1 receptor agonist activity that results in a positive inotropic effect on the heart at higher doses. Norepinephrine also may cause side effects as headache, blurred vision, chest pain ,nervousness, bradycardia or tachycardia.

ELIGIBILITY:
Inclusion Criteria:

1. The study will include 90 adult female patients, 45 in each group (between 18-35 years old).
2. patients of ASA physical status class I and class II.
3. patients scheduled for elective cesarean section under spinal anesthesia.

Exclusion Criteria:

1. Patient refusal.
2. Contraindication to spinal anesthesia .
3. Patients known allergic to Midodrine or Norepinephrine.
4. Patients with preexisting cardiovascular or cerebrovascular disease.
5. Patients with diabetes mellitus.
6. Patients with psychiatric disease or on psychiatric treatment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post spinal anesthesia hypotension | within 60 minutes of induction of spinal anesthesia
  decrease in Mean Arterial Blood Pressure more than 20% of the baseline reading

SECONDARY OUTCOMES:
Intraoperative ephedrine consumption | within 60 minutes of induction of spinal anesthesia
  ephedrine dose injected intravenous to control post spinal hypotension
Incidence of post spinal anesthesia bradycardia | within 60 minutes of induction of spinal anesthesia
  decrease in Heart Rate less than 50 Beats per minutes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCrae AF, Wildsmith JA. Prevention and treatment of hypotension during central neural block. Br J Anaesth. 1993 Jun;70(6):672-80. doi: 10.1093/bja/70.6.672. PMID 8329261
- [Background] Alseoudy MM, Nasr MO, Abdelsalam TA. Efficacy of Preoperative Oral Midodrine in Preventing Hypotension After Spinal Anesthesia in Young Adults: A Randomized Controlled Trial. Anesth Analg. 2022 Nov 1;135(5):1089-1096. doi: 10.1213/ANE.0000000000006173. Epub 2022 Aug 10. PMID 35950781
- [Background] Quaglia MG, Farina A, Palmery M, Desideri N, Donati E, Bossu E, Strano S. Chiral investigation of midodrine, a long-acting alpha-adrenergic stimulating agent. Chirality. 2004 Jul;16(6):356-62. doi: 10.1002/chir.20041. PMID 15190580
- [Background] Gutman LB, Wilson BJ. The Role of Midodrine for Hypotension Outside of the Intensive Care Unit. J Popul Ther Clin Pharmacol. 2017 Aug 23;24(3):e45-e50. doi: 10.22374/1710-6222.24.3.4. PMID 28873293